CLINICAL TRIAL: NCT03840941
Title: The Effect Of Frailty Level On Balance, Cognition And Activities Of Daily Living In COPD
Brief Title: The Effect of Frailty on Balance, Activities of Daily, and Exercise Capacity in COPD
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Deniz Inal-Ince, Prof. Dr., Hacettepe University
Other Study IDs: GO 18/83-22
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: COPD; Frailty
Keywords: COPD; Frailty; Balance; Cognition; Activities of Daily Living
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Frailty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frail patients with COPD: No intervention
- Non-frail patients with COPD: No intervention

SUMMARY:
The investigators aim to demonstrate whether balance, cognition and activities of daily living have changed in COPD patients with and without frailty.

DETAILED DESCRIPTION:
COPD is a common, preventable and treatable disease characterized by progressive respiratory symptoms and airflow limitation. Frailty defines a clinical syndrome characterized by multiple system effects, leading to decreased functional reserve and increased sensitivity to dependence or mortality following minor stress events. Inflammation, lack of physical activity, reduced exercise efficiency and maximum oxygen uptake may contribute to the development of frailty in patients with COPD. Balance, cognition and activities of daily living are associated with COPD.

This study will evaluate the effect of frailty on balance, cognition and activities of daily living in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients who have been clinically stable for the last four weeks and who have not undergone drug change for the last four weeks
* Being 55 years of age or older
* Accepted to participate in the study (Able and wililing to complete the informed consent process)
* Co-operate
* Patients with COPD who are ambulant without support or an assistive device

Exclusion Criteria:

* Neurological, cardiac or orthopedic diseases
* Other chronic diseases that may affect balance and walking

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who are diagnosed with COPD at Hacettepe University and who are referred to the Cardiopulmonary Rehabilitation Unit for physiotherapy also who are willing to participate in the study will be included in the study.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Presence of The Frailty Will Be evaluated Using The Frailty Criteria by Fried | 1st Day
  Frailty will be identified by the presence of three or more of the following criteria unintentional weight loss (10 Ibs in past year), weakness (grip strength), self-reported exhaustion, slow walking speed and low physical activity. Patients with three or more of the criteria present were classified as frail.
Balance Assessment Using Functional Reach Test | 1st Day
  The Functional Reach Test measures how far patient can reach forward from a normal relaxed stance.
Cognition Using MoCA-Test | 1st Day
  Cognitive function will be evaluated with the secreening tool the Montreal Cognitive Assessment (MoCA). The MoCA is a 30-point screening tool.
Perform activities of daily living (ADL) will be evaluated using the Glittre ADL-test | 1st Day
  Glittre ADL-test was designed specifically to assess the functional limitation in patients with COPD. Glittre ADL-test time will be considered the main outcome variable, and will be recorded in minutes (metric).

SECONDARY OUTCOMES:
Exercise Capacity Using 6-Minute Walk Test | 1st Day
  The standard protocol of the test is applied in a 30-meter continuous corridor. Standard instructions are given during testing.
Disease-Related Quality of Life Assessment | 1st Day
  COPD evaluation test (CAT) was developed to help assess health status.
Respiratory Muscle Strength Assessment | 1st Day
  Respiratory muscle strength will be evaluated by non-invasive methods by measuring maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP).
Shortness of Breath Assessment | 1st Day
  Modified Medical Research Council (mMRC) dyspnea scale will be used to determine the shortness of breath severity.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Inal-Ince, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Ankara, Sihhiye, Turkey (Türkiye)